CLINICAL TRIAL: NCT06490666
Title: The Change in Femoral Artery Pulsatility Index as a Novel Predictor to Post-spinal Hypotension in Adult Patient Undergoing Infraumbilical Surgeries, a Prospective Observational Study
Brief Title: (∆PI) to Predict Post-spinal Anesthesia Hypotension
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Adolf Helmy, Doctor, Cairo University
Other Study IDs: (∆PI) in spinal hypotension
Record Dates: First submitted 2024-06-29; First posted 2024-07-08 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Spinal Anesthesia Hypotension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: femoral artery doppler — femoral artery pulse wave doppler to measure both pulsatility and resistive indices

SUMMARY:
we aimed to evaluate the change in femoral artery pulsatility index as a predictor to post-spinal anesthesia hypotension

DETAILED DESCRIPTION:
After spinal anesthesia, hypotension is a common effect that occurs in between 15 and 30% of patients therefore it is essential to prevent such effect.

number of variables were utilized for estimating post spinal hypotension, such as assessing heart rate variability, perfusion index, inferior vena cava collapsibility index; however, the majority of these indices needs advanced equipment.

investigator of current research decided to study the role of ultrasound derived index namely pulsatility index to predict post spinal anesthesia hypotension.

ELIGIBILITY:
Inclusion Criteria:

* adult patient undergoing infra-umbilical surgeries.

Exclusion Criteria:

* coagulopathy peripheral vascular disease contraindication to spinal anesthesia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patient undergoing spinal anesthesia for infra-umbilical surgeries
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
change in pulsatility index to predict post spinal anesthesia induced hypotension | baseline and immediately after spinal anesthesia
  to measure PI before and after spinal anesthesia

SECONDARY OUTCOMES:
change in resistive index to predict post spinal anesthesia induced hypotension | baseline and immediately after spinal anesthesia
  to measure RI before and after spinal anesthesia
change in waveform morphology to predict post spinal hypotension | before and immediately after spinal anesthesia
  change of waveform morphology before and after spinal anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Hartmann B, Junger A, Klasen J, Benson M, Jost A, Banzhaf A, Hempelmann G. The incidence and risk factors for hypotension after spinal anesthesia induction: an analysis with automated data collection. Anesth Analg. 2002 Jun;94(6):1521-9, table of contents. doi: 10.1097/00000539-200206000-00027. PMID 12032019
- [Result] Wesselink EM, Kappen TH, Torn HM, Slooter AJC, van Klei WA. Intraoperative hypotension and the risk of postoperative adverse outcomes: a systematic review. Br J Anaesth. 2018 Oct;121(4):706-721. doi: 10.1016/j.bja.2018.04.036. Epub 2018 Jun 20. PMID 30236233
- [Result] Yu C, Gu J, Liao Z, Feng S. Prediction of spinal anesthesia-induced hypotension during elective cesarean section: a systematic review of prospective observational studies. Int J Obstet Anesth. 2021 Aug;47:103175. doi: 10.1016/j.ijoa.2021.103175. Epub 2021 May 1. PMID 34034957